CLINICAL TRIAL: NCT01468376
Title: An Open-label, Dose-finding Pilot Study of Various Formulations of Glucose-lowering Products in Otherwise Healthy Individuals With Impaired Glucose Tolerance
Brief Title: GLU-xx Formulations in Individuals With Impaired Glucose Tolerance
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor company was acquired and new owner chose not to proceed with clinical study
Sponsor: Afexa Life Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GLU-00-2010-1
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Impaired Glucose Tolerance
Keywords: impaired glucose tolerance; pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- GLU-01 (Experimental)
  Interventions: Dietary Supplement: GLU-01
- GLU-02 (Experimental)
  Interventions: Dietary Supplement: GLU-02
- GLU-03 (Experimental)
  Interventions: Dietary Supplement: GLU-03
- GLU-04 (Experimental)
  Interventions: Dietary Supplement: GLU-04
- GLU-05 (Experimental)
  Interventions: Dietary Supplement: GLU-05
- GLU-06 (Experimental)
  Interventions: Dietary Supplement: GLU-06

INTERVENTIONS:
Dietary Supplement: GLU-01 — 14 day dosing
  Arms: GLU-01
Dietary Supplement: GLU-02 — 14 day dosing
  Arms: GLU-02
Dietary Supplement: GLU-03 — 14 day dosing
  Arms: GLU-03
Dietary Supplement: GLU-04 — 14 day dosing
  Arms: GLU-04
Dietary Supplement: GLU-05 — 14 day dosing
  Arms: GLU-05
Dietary Supplement: GLU-06 — 14 day dosing
  Arms: GLU-06

SUMMARY:
The purpose of this study is to determine a safe,tolerable and efficacious dose of GLU-xx.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults between 21-65 years of age
* Body Mass Index (BMI) between 25 and ≤40
* OGTT (75g glucola) peak value between ≥140mg/dl and ≤199 mg/dl at screening visit
* Willingness to adhere to the requirements of the protocol, including availability for follow-up visits and donation of blood samples
* Willingness and ability to sign written informed consent
* Women of child bearing capacity who agree to use an acceptable form of birth control during the trial [i.e., oral contraception, reliable use of a double-barrier method (e.g., condom and diaphragm, condom and foam, condom and sponge), IUD or tubal ligation]

Exclusion Criteria:

* Active diabetes mellitus [fasting blood glucose of ≥7.0 mmol/L (≥126 mg/dL) or ≥11.1 mmol/L (≥200 mg/dL) after OGTT]
* Current coronary artery/ cardiovascular disease or history of a cardiovascular event (stroke, transient ischemic attack, myocardial infarction, angioplasty or coronary artery bypass grafting, angina pectoris) or have undergone a cardiovascular intervention within the past three months
* Seizure disorder
* Blood disorders, including anemia (i.e., hemoglobin levels less than 13 g/dL in men and less than 12 g/dL in women)
* Active infection, including HIV, hepatitis, etc
* Participants on Estrogen replacement must be on a stable dose for at least 3 months
* Serious illness requiring ongoing medical care or medication
* Gastrointestinal disorders or prior gastrointestinal surgeries (including gastric bypass or lap-band) that might cause complications or influence motility or satiety (e.g.,diverticulitis, inflammatory bowel disease, irritable bowel syndrome, intestinal narrowing or obstruction, difficulty swallowing)
* Any congenital spinal cord deformities or traumatic spinal cord injuries
* Uncorrected hypothyroidism
* Other significant metabolic endocrine disease
* Active liver disease or liver function impairment as evidenced by a history of liver disease or liver enzyme elevations >three times the upper limit of normal
* Current cancer
* Significant kidney disease (calculated by eGFR <60 mL/min)
* History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological,or psychiatric disorders which in the opinion of the investigator would be expected to interfere with the study or increase risk to the subject
* Use of anticoagulants such as warfarin
* Use of medications that might affect weight or food absorption (e.g., diuretics,glucocorticoids, anorexigenic agents, Orlistat, laxatives)
* Treatment within the previous 6 months with any medication that is known to affect glucose levels (such as insulin with or without an amylin analogue, sulfonylureas,meglitinides, biguanide metformin, thiazolidinediones, alpha-glucosidase inhibitors,oral dipeptidyl-peptidase-4 inhibitor, Sitagliptin, Incretin mimetic)
* Regular use of natural health products or dietary supplements known to affect glucose levels (such as chromium, zinc, fenugreek, cinnamon). If the participant agrees to stop taking these products 14 days prior to study entry and for the duration of the study, they can participate in the study

  o Any other natural health products or dietary supplements, with the exception of vitamins and minerals with dose of < 600 mg/day of vitamin E and containing no vitamin K. Natural health products or dietary supplements include products such as, but not limited to, Echinacea, Ginseng, St. John's Wort, Gingko, Glucosamine, Fish Oil supplements, Evening Primrose Oil, Green Tea or other herbal products consumed in the form of pills, extracts, capsules, or tablets. If the participant agrees to stop taking these products 14 days prior to study entry and for the duration of the study, they can participate in the study
* Vegan or Vegetarian
* Pregnant or lactating women, or intending to become pregnant
* Known allergy to any ingredient in the study product
* Any significant auto-immune disease

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Glucose and insulin response to the Oral Glucose Tolerance Test after administration of GLU-xx formulations | 14 days

SECONDARY OUTCOMES:
Safety and tolerability of GLU-xx formulations | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Jay Udani, MD, Principal Investigator — Medicus Research LLC/Staywell Research LLC
Locations (1):
- Staywell Research LLC, Northridge, California, United States